CLINICAL TRIAL: NCT02458872
Title: Impact of a Data-driven Monitor Alarm Reduction Strategy Implemented in Safety Huddles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Academic Pediatric Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-011896
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Hospitalization
Keywords: Clinical Alarms; Patient Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Safety huddle alarm intervention.
  Interventions: Behavioral: safety huddle alarm intervention
- Control Arm (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: safety huddle alarm intervention — The intervention consists of a monitor alarm dashboard that displays the numbers and types of alarms for each patient, and an accompanying checklist to guide data-driven discussion of 2-4 patients with high alarm rates.
  Arms: Intervention Arm

SUMMARY:
This is a pragmatic, paired, cluster-randomized controlled trial evaluating the impact of a safety huddle-based intervention on physiologic monitor alarm rates on pediatric inpatient units.

DETAILED DESCRIPTION:
Hospital physiologic monitors can alert clinicians to early signs of physiologic deterioration, and thus have great potential to be life-saving. However, monitors generate frequent alarms, most of which are non-actionable.

When clinicians become overburdened with alarms, they begin to exhibit alarm fatigue: responding more slowly to alarms or ignoring alarms entirely. In this protocol the investigators outline the methods they will use to evaluate the impact of a safety huddle-based intervention on physiologic monitor alarm rates using a pragmatic, paired, cluster-randomized controlled trial with the intervention delivered at the unit level. This work is considered quality improvement research, and some of the approaches described in this protocol are from the field of quality improvement.

Currently, at most hospitals data like this on the numbers of alarms that patients generate are only available to researchers with the software tools needed to interrogate and record data from the monitor network. The goal of this proposal is to bring this data to the safety huddles occurring daily on inpatient units in an accessible format to help teams make informed decisions about monitoring and minimize the potential of harm from alarm fatigue.

ELIGIBILITY:
Inclusion criteria: Any nurse, physician, nurse practitioner, or physician assistant caring for a patient whose alarms are discussed in a safety huddle on an intervention unit.

Exclusion criteria: none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77280 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the unit-wide rate of alarms per patient-day at 44 weeks | Baseline and 44 weeks

SECONDARY OUTCOMES:
Pre-post huddle patient-level difference in differences of alarm rates | The 24 hours before a safety huddle opportunity versus the 24 hours before a safety huddle opportunity
  The difference in the rate of alarms in individual patients in the 24 hours after discussion in a huddle compared with themselves in the 24 hours before the huddle, patients on the same unit as the huddle but whose alarms are not discussed, and patients on units without the alarm huddle intervention.
Implementation outcomes | Within 4 hours after the huddle intervention occurred
  Proportion of huddles in post-implementation data collection period that included discussion of at least 1 patient's alarms, proportion of patients in whom a change in monitor delay time was recommended who had delay time changed in a direction consistent with the recommendations within 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Bonafide, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bonafide CP, Localio AR, Sternler S, Ahumada L, Dewan M, Ely E, Keren R. Safety Huddle Intervention for Reducing Physiologic Monitor Alarms: A Hybrid Effectiveness-Implementation Cluster Randomized Trial. J Hosp Med. 2018 Sep 1;13(9):609-615. doi: 10.12788/jhm.2956. Epub 2018 Feb 27. PMID 29489921